CLINICAL TRIAL: NCT07237412
Title: Neurofeedback-based Visual Restoration Therapy
Acronym: ReViseNetFeed
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adrian Guggisberg (Other)
Responsible Party: Sponsor-Investigator, Adrian Guggisberg, Full Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-00765
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Visual Field Defect Homonymous Bilateral
Keywords: stroke; neurofeedback; network; EEG
MeSH Terms: conditions — Hemianopsia; Stroke | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active phase (Active Comparator): During the active phase, patients will receive real-time audio feedback on spontaneous alpha-band functional connectivity between ipsilesional associative visual areas and the rest of the brain. This will allow them to learn to improve their pathological brain interactions. The neurofeedback training will last about 40 minutes, with frequent breaks. It will be followed by visual stimulation of the affected visual field according to recommendations for inducing steady-state visual evoked potentials.
  Interventions: Procedure: neurofeedback
- control phase (Sham Comparator): The control phase is structured identically to the active period, except that the acoustic neurofeedback is synthetically generated and not linked to the subject's actual functional connectivity, while still resembling its dynamic characteristics to ensure effective blinding. The training will last about 40 minutes, with frequent breaks. The training will be followed by visual stimulation of the affected visual field, just as in the active condition.
  Interventions: Procedure: neurofeedback

INTERVENTIONS:
Procedure: neurofeedback — The proposed neurofeedback approach relies on high-density electroencephalography (EEG) combined with advanced source localization algorithms. Data will be analyzed in real-time and simultaneously recorded for offline analysis. During each update, a data segment will be filtered between 1 and 20 Hz. The beamformer, computed at the beginning of the session, will be used to project the signal to the gray-matter voxels.
  The investigators will compute the alpha-band absolute imaginary coherence between a visual target area and the rest of the brain as index of functional connectivity. Global functional connectivity in the alpha band (8-13 Hz) between the voxels in the target region and the rest of the brain will be calculated.

SUMMARY:
Visual field defects are a common consequence of acquired brain injuries and affect people of all ages. These vision problems make everyday life more difficult-for example, when reading, driving, or moving around safely. However, there is currently no effective therapy to improve visual field defects.

Previous training methods have focused on maximizing brain activity during a task. However, new findings show that the best performance is achieved when the brain is already in a state of high communication before the task. Our research shows that people can learn to increase communication between brain regions through neurofeedback.

Studies have shown that neurofeedback can help people after a stroke: it improves the coordination of brain areas that are important for movement, thereby helping to increase mobility. Building on these findings, this study investigates whether EEG neurofeedback can support the visual centers in the brain to improve vision in patients with chronic visual field defects. The main objective of the study is to evaluate the effectiveness of neurofeedback in improving visual field defects. More specifically, the investigators are investigating the development of visual ability (expansion of the visual field, contrast sensitivity).

ELIGIBILITY:
Inclusion Criteria:

* Chronic, stable HVFD (homologous lateral quadranopsia or hemianopsia)
* 12 months or more after stroke
* Age range 50-70
* Ability to provide informed consent

Exclusion Criteria:

* Inability to concentrate for long treatment sessions
* Eye disease with impact on visual field or acuity
* Presence of non-MRI safe metal in the body
* New stroke during study period
* Hemispatial neglect

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual field | Change from enrollment to post-test at 3 weeks and follow up at 7 weeks (repeated-measures ANOVA)
  This will be evaluated using the Haag-Streit Octopus 900 perimetry device (Haag-Streit AG, Köniz, Switzerland). The device features advanced gaze-tracking capabilities that effectively control compensatory eye movements, ensuring accurate measurement of visual field improvements. The Central 30-2 protocol will be followed.
  The primary outcome will be the change in the Mean Deviation (MD) score in detection threshold (in dB) from baseline to the end of the intervention period within the target area of affected visual field. The MD score represents the overall deviation of the patient's visual field from age-matched normative data, with more negative values indicating greater visual field loss.

SECONDARY OUTCOMES:
Changes in alpha-band functional connecticity | Change from entrollment to the end of treatment at 3 weeks.
  Neurophysiological changes reflected in alpha-band network communication between targeted area and the rest of the brain, as measured with EEG-based FC. For this, the investigators will record resting state EEG, which, together with individual MRI scans and beamforming techniques, will allow us to estimate FC in source space.
Questionnaire on daily-life impact of the visual impairment | Change from enrollment to treatment end at 3 weeks
  Daily-life impact of the visual impairment (visual function questionnaire, VFQ25). It ranges from 0 (worst visual function) to 100 (best visual function)).
Reading speed | Change from enrollment to treatment end at 3 weeks and follow up at 7 weeks (repeated-measures ANOVA).
  Reading speed (International Reading Speed Test, IReST). It is a continuous variable measured in words per minute with no predefined scale range (higher values indicate better performance).

OTHER OUTCOMES:
Test of Attentional Performance (TAP) Visual Scanning | Change from enrollment to treatment end at 3 weeks
  Reaction time in the TAP Visual Scanning test is a continuous variable with no predefined bounds, with longer reaction times indicating poorer performance; omissions represent the number of missed targets, with higher values also indicating poorer performance.
Test of Attentional Performance (TAP) Sustained Attention | Change from enrollment to treatment end at 3 weeks.
  The reaction time of the TAP Sustained Attention is a continuous variable with no predefined bounds, with longer reaction times indicating poorer performance; omissions represent the number of missed targets, with higher values also indicating poorer performance.
Test of Attentional Performance (TAP) Visual field and Neglect test | Change from enrollment to treatment at 3 weeks.
  The reaction time is a continuous variable with no predefined bounds, with longer reaction times indicating poorer performance; omissions represent the number of missed targets, with higher values also indicating poorer performance.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Inselspital, Bern, Canton of Bern
  - Division of Neurorehabilitation, University Hospital of Geneva, Geneva, Canton of Geneva

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sabel BA, Henrich-Noack P, Fedorov A, Gall C. Vision restoration after brain and retina damage: the "residual vision activation theory". Prog Brain Res. 2011;192:199-262. doi: 10.1016/B978-0-444-53355-5.00013-0. PMID 21763527
- [Background] Mottaz A, Corbet T, Doganci N, Magnin C, Nicolo P, Schnider A, Guggisberg AG. Modulating functional connectivity after stroke with neurofeedback: Effect on motor deficits in a controlled cross-over study. Neuroimage Clin. 2018 Jul 30;20:336-346. doi: 10.1016/j.nicl.2018.07.029. eCollection 2018. PMID 30112275
- [Background] Allaman L, Mottaz A, Kleinschmidt A, Guggisberg AG. Spontaneous Network Coupling Enables Efficient Task Performance without Local Task-Induced Activations. J Neurosci. 2020 Dec 9;40(50):9663-9675. doi: 10.1523/JNEUROSCI.1166-20.2020. Epub 2020 Nov 6. PMID 33158966
- [Background] Allaman L, Mottaz A, Guggisberg AG. Disrupted resting-state EEG alpha-band interactions as a novel marker for the severity of visual field deficits after brain lesion. Clin Neurophysiol. 2021 Sep;132(9):2101-2109. doi: 10.1016/j.clinph.2021.05.029. Epub 2021 Jun 28. PMID 34284245